CLINICAL TRIAL: NCT01863342
Title: Influence of Central Sensitization on Efficacy of Patient-controlled Epidural Analgesia in Osteoarthritis Patients Undergoing Total Knee Replacement
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2013-0127
Record Dates: First submitted 2013-05-22; First posted 2013-05-27 (Estimated); Last update posted 2013-05-27 (Estimated); Status verified 2013-05

CONDITIONS: Knee Osteoarthritis
Keywords: central sensitization; osteoarthritis; epidural analgesia
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- CSI score < 40: CSI cutoff value<40
  Interventions: Procedure: CSI score < 40
- Group 2: CSI score ≥ 40: CSI cutoff value≥40
  Interventions: Procedure: CSI score ≥ 40

INTERVENTIONS:
Procedure: CSI score < 40
  Groups: CSI score < 40
Procedure: CSI score ≥ 40
  Groups: Group 2: CSI score ≥ 40

SUMMARY:
Nociceptor inputs can trigger a prolonged but reversible increase in the excitability and synaptic efficacy of neurons in central nociceptive pathways, the phenomenon of central sensitization. The degenerative joint disease, osteoarthritis, with characteristic destruction of cartilage and alteration in bone is a very common cause of chronic pain. The degree of pain does not always correlate with the extent of joint damage or presence of active inflammation raising the possibility that there may be a central component to the pain. The central sensitization inventory (CSI) is a new self-report screening instrument to measure the degree of central sensitization, and to help identify patients with central sensitivity syndromes. The aim of this investigation is to evaluate the influence of preoperative central sensitization, which represented by CSI score, on postoperative pain score in osteoarthritis patients undergoing total knee replacement who receiving patient-controlled epidural analgesia.

ELIGIBILITY:
Inclusion Criteria:

* Aged 20 to 80 years osteoarthritis patients undergoing total knee replacement under spinal anesthesia, and who receiving postoperative epidural PCA

Exclusion Criteria:

* refusal
* coagulopathy
* neurologic deficit
* preoperative opioids medication
* recent analgesics change

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: osteoarthritis patients undergoing total knee replacement
Sampling Method: Non-Probability Sample
Enrollment: 98 (Estimated)
Dates: Start 2013-05; Primary Completion 2014-05 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Peak pain score | at the point of Epidural PCA to postoperative 1-48 h
  Numeric rating scale (0 to 10 points) at each assessment interval

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Yonsei University College of Medicine, Seoul, Seoul, South Korea